CLINICAL TRIAL: NCT04585386
Title: Pilot Study to Assess the Efficacy of the ATLAS Medical Device on Pain in Patients With Subacute or Chronic Low Back Pain With Lumbar Disc Disease: Prospective, Randomized Trial (AmbuTract)
Brief Title: Efficacy of the ATLAS Medical Device on Pain in Patients With Low Back Pain Due to Lumbar Disc Disease
Acronym: AmbuTract
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision: no sufficient patient
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A01625-34
Record Dates: First submitted 2020-10-12; First posted 2020-10-14 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Lumbar Disc Disease
MeSH Terms: conditions — Intervertebral disc disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATLAS (Experimental): Medical device named ATLAS which is an "active corset" (rigid lumbar restraint) and connected.
  Interventions: Other: Visual analog scale; Other: Mac Gill Pain Questionnaire; Other: Roland and Morris Disability Questionnaire; Other: Quebec questionnaire
- Standard lumbar support belt (Active Comparator): Standard lumbar support belt : LombaSkin® or Lombogib®
  Interventions: Other: Visual analog scale; Other: Mac Gill Pain Questionnaire; Other: Roland and Morris Disability Questionnaire; Other: Quebec questionnaire

INTERVENTIONS:
Other: Visual analog scale — to measure the lumbar and radicular pain felt by the patient.
Other: Mac Gill Pain Questionnaire — self-questionnaire that allows a qualitative assessment of chronic pain
Other: Roland and Morris Disability Questionnaire — functional disability scale for assessing low back pain
Other: Quebec questionnaire — To access the patient's perception of incapacity

SUMMARY:
Monocentric, comparative, randomized, controlled interventionnal study in 2 parallel groups, aiming to compare the efficacy of the ATLAS device with that of a standard lumbar belt on the reduction of pain felt in patients with subacute or chronic low back pain with lumbar disc disease.

DETAILED DESCRIPTION:
The main expected benefit is a reduction in pain experienced in patients with subacute or chronic low back pain during and after wear. Consequently, an improvement in the quality of daily life is expected with a less significant impact of low back pain.

The main objective of the study is to compare the efficacy of the ATLAS medical device with a standard lumbar support belt in terms of immediate reduction of low back pain experienced in patients with subacute or chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from subacute (for 6 to 12 weeks) or chronic (> 3 months) lumbar pain;
* Lumbar disc disease confirmed by Magnetic Resonance Imaging (MRI) less than 3 months old;
* Patient with lumbar pain ≥ 40mm on the visual analogue scale (VAS) at inclusion;
* Patient in whom a lumbar belt / restraint is considered for a short period to help resumption of activity;
* Patient with internet and a camera (by phone or computer) and agreeing to use them as part of the study's teleconsultations;
* Patient capable of understanding the information related to the study (absence of linguistic, psychological, cognitive problem, etc.), of reading the information leaflet, of completing questionnaires and agreeing to sign the consent form.

Exclusion Criteria:

* Patient with neurological radicular or medullary deficits;
* Patient presenting a postural problem with lateralized contracture;
* Skin pathology in the trunk region and / or contusions and injuries by stretching the trunk;
* History of spinal arthrodesis surgery;
* History of cauda equina syndrome;
* Patient treated by implanted neurostimulation;
* Scoliosis with Cobb angle> 30 °;
* History of recent fracture of the dorsolumbar spine (<3 months);
* History of recent rib fracture (<3 months);
* History of recent herniated disc surgery (<3 months);
* Patient with diagnosed fracture osteoporosis;
* Patient with heart or circulatory disease or respiratory failure;
* Patient presenting with a tumor or infectious process of the vertebrae;
* Pregnant or likely to be (of childbearing age, without effective contraception) or breastfeeding;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Patient not beneficiary of a social security scheme.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Evolution of the lumbar pain | 1 hour after the start of the port
  The primary outcome measure is the change in lumbar pain assessed by the patient using an VAS from 0 to 100 mm.

SECONDARY OUTCOMES:
To assess the safety and tolerance of the devices | Between Day 0 and Day 8
  Analysis of all adverse events collected during the study
Satisfaction of the patient | After a period of 8 days of wearing the medical device
  Percentage of patients with an overall assessment of the device

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Le Bois, Lille, France

IPD SHARING:
Plan to Share IPD: No